CLINICAL TRIAL: NCT05677984
Title: Comparison the Prescription of Duration of Awaken Prone Positioning Ventilation Duration in COVID-19 Patients: a Randomised Controlled Study
Brief Title: Awaken Prone Positioning Ventinlation in COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Professor, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20221227
Record Dates: First submitted 2023-01-03; First posted 2023-01-10 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APP group (Experimental): Directive APP for a target of 12 hours per day or more
  Interventions: Procedure: Awaken prone positioning ventilation
- Control group (No Intervention): No intervention on APP

INTERVENTIONS:
Procedure: Awaken prone positioning ventilation — patients were mandated to keep a prone position for at least 12 hours.
  Arms: APP group

SUMMARY:
Awaken prone positioning (APP) ventilation has been widely accepted as a standard regimen in the management of COVID-19 patients. Physiological studies have proved ventilation/perfusion improvement during APP in COVID-19, which was associated improved oxygenation. However, the optimal duration for APP was not yet demonstrated. In this study, we aimed at the prolonged APP to see whether this could improve patients outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 18-yr to 85-yr
* Severe COVID-19 pneumonia (with typical radiographic alternations) and non-intubated patients.
* SpO2 <= 93% with ambient air at rest.
* PaO2/FiO2 <= 300 mmHg

Exclusion Criteria:

* Definite intolerance to APP (e.g. pregnancy, extremity deformity, recent fracture, open thoracic or abdominal surgery, pace-maker implant in recent 48-hr, spine stability, pelvis or facial fractures, predicted difficult airway)
* morbidity obesity, BMI > 40
* consciousness disorder (GCS < 13), delirium dementia
* hemodynamic instability (with norepinephrine >20 ug/min )
* NYHA Grade III or IV
* Severe hemoptysis
* long term home oxygenation of CPAP
* Refuse invasive mechanical ventilation (DNI DNR)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
28-day intubation rate | follow-up till 28-day
  whether the patients' were intubated

SECONDARY OUTCOMES:
APP duration/days | follow-up till APP ended, daily duration of APP also recoreded, up to 7 days
  hours of APP per day
Application of HFNC NIV vasopressor CRRT ECMO sedation, or complication | follow-up till 28-day
  Whether to apply these treatments，any complications occur,days free from respiratory support and days free from invasive mechanical ventilation at 28 day
mortality (ICU hospital) length of ICU (hospital) stay | follow-up during the ICU/hospital stay, up to 28 days
  mortality AND mortality and length of stay at 28 day

OTHER OUTCOMES:
Adverse events of interest | 28 post-randomisation
  All adverse events of interest that occur in both randomised arms will be reported up to day 28 post-randomisation, including the following:
  * Nausea,
  * Unintentional removal of intravenous access,
  * Pressure ulcer,
  * Unexpected respiratory cardiac arrest Nausea, Unintentional removal of intravenous access, Pressure ulcer，Unexpected respiratory cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Haibo QIU, Dr, Study Director — Southeast University
Locations (1):
- Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
from the email：liulingdoctor@126.com
Time Frame: Starting from the official publication of the manuscript to 1 year later
Access Criteria: collaborator

REFERENCES:
- [Derived] Sun Q, Zhang R, Zhang J, Xie J, Huang Y, Yang Y, Qiu H, Liu L, Chen H; Chi-ARDS Net (Chinese ARDS Research Network). Impact of awake prone positioning duration on intubation or mortality in COVID-19 patients with acute respiratory failure: secondary analysis of a randomized clinical trial. Ann Intensive Care. 2025 Jun 23;15(1):84. doi: 10.1186/s13613-025-01501-8. PMID 40549277
- [Derived] Liu L, Sun Q, Zhao H, Liu W, Pu X, Han J, Yu J, Jin J, Chao Y, Wang S, Liu Y, Wu B, Zhu Y, Li Y, Chang W, Chen T, Xie J, Yang Y, Qiu H, Slutsky A; Chi-ARDS Net (Chinese ARDS Research Network). Prolonged vs shorter awake prone positioning for COVID-19 patients with acute respiratory failure: a multicenter, randomised controlled trial. Intensive Care Med. 2024 Aug;50(8):1298-1309. doi: 10.1007/s00134-024-07545-x. Epub 2024 Aug 1. PMID 39088076